CLINICAL TRIAL: NCT06568783
Title: Evaluation of Patients With Refractory Dermatomyositis Using [18F]- Fibroblast Activation Protein Inhibitor-74 (FAPI-74) PET/MRI Imaging
Brief Title: Evaluation of Patients With Refractory Dermatomyositis Using [18F] FAPI-74 PET/MRI Imaging
Acronym: FAPI-74
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Farshad Moradi (Other)
Responsible Party: Sponsor-Investigator, Farshad Moradi, Clinical Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74917
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Refractory Dermatomyostitis

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm study enrolling 21 adult participants to evaluate [18F]-FAPI-74 PET/ MRI for assessment of muscle and soft tissue involvement in Dermatomyositis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]-FAPI-74 PET/ MRI (Experimental): Participant receive [18F]-FAPI-74 injection and approximately 45-60 minutes later receive a MRI scan from vertex to legs, followed by a static PET emission scan over the same area.
  Interventions: Drug: [18F]-FAPI-74

INTERVENTIONS:
Drug: [18F]-FAPI-74 — [18F]-FAPI-74 7 mCi ± 20% administered intravenously.

SUMMARY:
This study proposes the use of a PET isotope, [18F]-Fibroblast Activation Protein Inhibitor-74, for a prospective single-center, single-arm study using MRI imaging for participants with Refractory Dermatomyostitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected dermatomyositis.
2. Patient must be > 18 years old.
3. Be willing and able to provide written informed consent for the trial.

Exclusion Criteria:

1. Women who are pregnant or potentially pregnant per the Department of Radiology Policy on Imaging in Potentially Pregnant and Pregnant Women.
2. Contraindication to MRI or inability to lie flat for 30 min
3. Any serious medical condition that in the opinion of principal investigator could pose significant risk of harm or injury to the patient if they participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Rate of [18F]-FAPI-74 uptake. | up to 1 hour
  write the outcome title, how it will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share.

REFERENCES:
- [Background] Bergmann C, Distler JHW, Treutlein C, Tascilar K, Muller AT, Atzinger A, Matei AE, Knitza J, Gyorfi AH, Luck A, Dees C, Soare A, Ramming A, Schonau V, Distler O, Prante O, Ritt P, Gotz TI, Kohner M, Cordes M, Bauerle T, Kuwert T, Schett G, Schmidkonz C. 68Ga-FAPI-04 PET-CT for molecular assessment of fibroblast activation and risk evaluation in systemic sclerosis-associated interstitial lung disease: a single-centre, pilot study. Lancet Rheumatol. 2021 Mar;3(3):e185-e194. doi: 10.1016/S2665-9913(20)30421-5. Epub 2021 Jan 25. PMID 38279381
- [Background] Giesel FL, Adeberg S, Syed M, Lindner T, Jimenez-Franco LD, Mavriopoulou E, Staudinger F, Tonndorf-Martini E, Regnery S, Rieken S, El Shafie R, Rohrich M, Flechsig P, Kluge A, Altmann A, Debus J, Haberkorn U, Kratochwil C. FAPI-74 PET/CT Using Either 18F-AlF or Cold-Kit 68Ga Labeling: Biodistribution, Radiation Dosimetry, and Tumor Delineation in Lung Cancer Patients. J Nucl Med. 2021 Feb;62(2):201-207. doi: 10.2967/jnumed.120.245084. Epub 2020 Jun 26. PMID 32591493
- [Background] Kuwert T, Schmidkonz C, Prante O, Schett G, Ramming A. FAPI PET Opens a New Window to Understanding Immune-Mediated Inflammatory Diseases. J Nucl Med. 2022 Aug;63(8):1136-1137. doi: 10.2967/jnumed.122.263922. Epub 2022 Apr 7. No abstract available. PMID 35393350
- [Background] Li J, Wei W, Xu W, Wu W, Liu J, Ye S. [68Ga]Ga-FAPI-04 and [18F]FDG PET/ CT in a patient with MDA5 dermatomyositis. Eur J Nucl Med Mol Imaging. 2023 Oct;50(12):3790-3791. doi: 10.1007/s00259-023-06291-4. Epub 2023 Jun 5. No abstract available. PMID 37272957
- [Background] Meyer C, Dahlbom M, Lindner T, Vauclin S, Mona C, Slavik R, Czernin J, Haberkorn U, Calais J. Radiation Dosimetry and Biodistribution of 68Ga-FAPI-46 PET Imaging in Cancer Patients. J Nucl Med. 2020 Aug;61(8):1171-1177. doi: 10.2967/jnumed.119.236786. Epub 2019 Dec 13. PMID 31836685
- [Background] Treutlein C, Distler JHW, Tascilar K, Fakhouri SC, Gyorfi AH, Atzinger A, Matei AE, Dees C, Buttner-Herold M, Kuwert T, Prante O, Bauerle T, Uder M, Schett G, Schmidkonz C, Bergmann C. Assessment of myocardial fibrosis in patients with systemic sclerosis using [68Ga]Ga-FAPI-04-PET-CT. Eur J Nucl Med Mol Imaging. 2023 May;50(6):1629-1635. doi: 10.1007/s00259-022-06081-4. Epub 2022 Dec 16. PMID 36522438
- [Background] Wu J, Qiu L, Wang Y, Zhang C. Dermatomyositis on 68Ga-FAPI PET/CT in a Patient With Nasopharyngeal Carcinoma. Clin Nucl Med. 2022 Feb 1;47(2):149-150. doi: 10.1097/RLU.0000000000003809. PMID 34284484
- [Background] Zheng J, Chen H, Lin K, Yao S, Miao W. [68Ga]Ga-FAPI and [18F]FDG PET/CT images in a patient with juvenile polymyositis. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):2051-2052. doi: 10.1007/s00259-020-05185-z. Epub 2021 Jan 18. No abstract available. PMID 33462628